CLINICAL TRIAL: NCT07078058
Title: Low Level Laser Versus Transcutaneous Vagus Nerve Stimulation on Vascular Changes in Patients With Diabetic Polyneuropathy
Brief Title: Low Level Laser VS Transcutaneous Vagus Nerve Stimulation on Vascular Changes in Patients With Diabetic Polyneuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Manar Elbaz, Principal Investigator, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manar-005515
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Low Level Laser; Transcutaneous Vagus Nerve Stimulation; Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser (Experimental): Patients will receive Low Level Laser irradiated with two wavelengths of visible 630 nm and near infra-red 810 nm for 15 min on entire surface of each foot three times a week for 2 months
  Interventions: Device: Low level laser
- Transcutaneous auricular Vagus nerve stimulation (Active Comparator): Patients will receive 30 minutes Transcutaneous auricular Vagus nerve stimulation 5 sessions per week for 2 months.
  Interventions: Device: Transcutaneous auricular Vagus nerve stimulation

INTERVENTIONS:
Device: Low level laser — Patients in the low level laser group will be irradiated with visible and near-infra-red lasers at a pulsed mode with a frequency of 35 Hz, peak power of 100 mW, and a spot diameter of 5 mm. The 15-minute sessions were performed three times a week for two months, with each laser having a power density of 0.35 mW/cm2 and an energy density of 32.08 J/cm2.
  Arms: Low Level Laser
Device: Transcutaneous auricular Vagus nerve stimulation — Patients will receive 30 minutes of transcutaneous vagus nerve stimulation for 2 months, with 5 sessions per week. The antihelix and cymba concha will be sterilized with 75% alcohol, and the electrode will be attached. The device parameters include a wave width of 0.2 ms ± 30%, pulse frequency of 20 Hz, gradually increasing intensity to a tolerable intensity (4-6 mA), and duration of 30 minutes.
  Arms: Transcutaneous auricular Vagus nerve stimulation

SUMMARY:
To compare the effect of both low-level laser versus transcutaneous vagus nerve stimulation on vascular changes in patients with diabetic polyneuropathy

DETAILED DESCRIPTION:
Diabetic polyneuropathy is a prevalent and severe diabetes-related complication linked to cardiovascular mortality and disease events, even after accounting for risk factors and diabetes status.

Diabetic polyneuropathy affects the peripheral nervous system, leading to dysfunctions in sensory, motor, and autonomic nervous systems. It predisposes diabetics to refractory neuropathic pain, foot ulcers, and amputation, lowering quality of life, increasing mortality, and prompting patients with diabetes to seek medical attention.

Over half of diabetes patients experienced painful diabetic polyneuropathy over the past few decades Painful diabetic polyneuropathy therapy uses various drugs for symptom relief, but they often have systemic side effects and do not slow neuropathy progression. Therefore, investigating non-pharmacological interventions like low-level laser and transcutaneous auricular vagus nerve stimulation is crucial for developing more effective and potentially safer pain management options.

low-level laser therapy and transcutaneous auricular vagus nerve stimulation are emerging non-invasive interventions that have shown potential in alleviating pain associated with diabetic polyneuropathy, a common diabetes complication affecting quality of life.

The effectiveness of conservative treatment options for painful diabetic polyneuropathy needs further investigation. If one method proves superior in reducing pain, improving macrovascular health, and quality of life, it could guide clinical decisions

ELIGIBILITY:
Inclusion Criteria:

The patient selection will be according to the following criteria:

1. 30 patients diagnosed with diabetic neuropathy from both genders their ages will be ranged from 45-60 years old.
2. All patients are ambulant independently.
3. All patients are under full medical control
4. Glycated hemoglobin is ranged from 6.5: 7 %.
5. Patients have had diabetes for more than 5 or 10 years.
6. patients experiencing painful peripheral neuropathic symptoms for more than 6 months involving both lower extremities and complained of burning pain with paresthesia in both legs.

7 Neurological examination revealed abnormal sensation appeared at the ends of the extremities.

Exclusion Criteria:

1. Patients had unstable glycemic control and/or medical conditions that would confound assessment of neuropathy such as malignancy, active/untreated thyroid disease, peripheral vascular diseases, vascular insufficiency (claudication, skin discoloration, ulceration).
2. Following the implantation of cardiac pacemakers or other electrical stimulation devices.
3. Patient had sinus bradycardia, long QT syndrome, or other arrhythmias or mental disorders.
4. Patients whose heart rate dropped below 50 beats/min after vagus nerve stimulation.
5. Nerve damage as a result of prior reconstructive or replacement knee surgery, back surgery, spinal stenosis, spinal compression or radiculopathy

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
assessment of change of vascular blood flow | at baseline and after 8 weeks
  The study uses Duplex Doppler ultrasound to assess vascular changes in the posterior tibial, anterior tibial, and peroneal arteries, assessing blood flow, Tunica intima thickness, and Resistive index using a variable frequency range.

SECONDARY OUTCOMES:
Assessment of change of Neuropathic Pain | at baseline and after 8 weeks
  The Douleur Neuropathique en 4 (DN4) is a screening questionnaire that consists of interview questions and physical tests to identify possible neuropathic pain. It has high test-retest and inter-rater reliability, with an ICC of 0.8 and a Cohen's kappa of 0.8. A total score is calculated as the sum of the 10 items. Scores _ 4 out 10 of indicate that neuropathic pain is likely.
Assessment of change of Quality of life | at baseline and after 8 weeks
  is a validated, comprehensive, self-administered questionnaire designed to measure the relationship between symptomatic DN and QOL from the perspective of the patient. The study used the Norfolk QOL-DN scoring algorithm to assess the quality of life of individuals. All symptom domain items were assigned a score, with items 31 and 32 scored on a 5-point Likert scale. Items 31 and 32 were scored on a scale of -2 to 2, with -2 indicating "Much Better" and -1 indicating "Somewhat Better." The summation of scores was based on total quality of life, physical functioning/large fiber, ADLs, symptoms, small fiber, and autonomic. A higher score on the Norfolk QOL-DN indicates a poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Horus university, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: No